CLINICAL TRIAL: NCT03607864
Title: Evaluation of Marginal Bone Loss After Immediate Implant Placement in Maxillary Esthetic Zone With Coral Bone Versus Xenograft
Brief Title: Coral Bone Graft Verses Xenograft With Immediate Implant in Maxillary Anterior Esthetic Zone
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: because bone osteointegration is completed
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amro Abdelaal Abdelhakim Elbahkiri, principal investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CairoUimplant
Record Dates: First submitted 2018-06-20; First posted 2018-07-31 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Badly Decayed Anterior Maxillary Teeth
MeSH Terms: interventions — Transplantation, Heterologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- coral bone graft and xenograft (Experimental): Extraction of upper anterior badly broken teeth with immediate implant placement with the use of coral bone and xenograft as grafting material between the implant and the labial socket bone
  Interventions: Device: coral bone graft and xenograft

INTERVENTIONS:
Device: coral bone graft and xenograft — ligible patients will be randomized in equal proportions between control group(immediate implant placement with grafting with xenograft) and study group (immediate implant placement with grafting with coral bone) Patients of both groups will be subjected to standard panoramic radiographs, cone beam ct .
  Crestal bone level will measured by cone beam ct. Local anesthesia will be given to the patient. Only sulcular incision line with reflection is used A peritome will be used for a traumatic extraction of remaining roots. The extraction socket will be evaluated for absence of any fenestration or granulation tissues implant will be inserted in extraction socket bodily palatal with grafting with coral bone and xenograft The flap will then be copiously irrigated with saline in preparation for closure.
  The flap will then be closed using interrupted 5/0 prolene sutures.

SUMMARY:
Autogenous bone graft is considered to be the golden standard for grafting as it has osteoconductive , osteoinductive and osteogenic functions , however it has the problems of donor site morbidity , the need for two surgeries as well as post operative swelling and discomfort of the patient , so alternative bone grafts as alloplast has been introduced.

Coral bone has a structure which is similar to that of cancellous bone , its mechanical properties is similar to that of bone and it consists of high content of calcium carbonate scaffolds that has the advantages of being biodegradable , biocompatible and osteoconductive , they act as a carrier for growth factors and allow cell attachment , growth , spreading , differentiation and has been found to be effective bone graft

DETAILED DESCRIPTION:
Immediate implant placement has the advantages of better esthetics , reduction in the number of surgeries (one surgery is needed) and reduction in the time of treatment so it is more suitable and comfortable for patients .

Immediate implant placement in fresh extraction socket after tooth extraction may reduce the incidence of bone loss compared to implant placement in the healed bone.

Certain studies showed that bone resorption occurs with immediate implant placement and there is high risk of failure and complications.

The gold standard for immediate implant placement is placing bone graft around the implant to fill the jumping gap between the implant and the socket.

Certain studies showed that if the jumping gap is 1-2 mm so no grafting is needed , but if the gap is more than 2mm then bone grafting is needed .

Immediate implant placement has the disadvantage of ; difficulty in obtaining primary stability , lack of adequate soft tissue coverage and also the control of the implant position is difficult in addition to the cost of the graft.

Despite these disadvantages the success rates of immediate implants is very high.

Autogenous bone graft is considered to be the golden standard for grafting as it has osteoconductive , osteoinductive and osteogenic functions , however it has the problems of donor site morbidity , the need for two surgeries as well as post operative swelling and discomfort of the patient , so alternative bone grafts as alloplast has been introduced.

Coral bone has a structure which is similar to that of cancellous bone , its mechanical properties is similar to that of bone and it consists of high content of calcium carbonate scaffolds that has the advantages of being biodegradable , biocompatible and osteoconductive , they act as a carrier for growth factors and allow cell attachment , growth , spreading , differentiation and has been found to be effective bone graft.

Certain studies showed that coral bone has similar results as autogenous bone and that it is encouraging for the osteoregenerative process resulting in tissue organization that allows for mechanical stability and function which is similar to that of native bone.

6b. Choice of the comparator: Xenografts are one of the most successful and widely used grafting materials nowadays as a replacement for autogenous bone grafts.

Studies showed that xenografts are very successful because of their osteoconductive properties , their denisty which provides stabilization to the graft and implant and they supply the necessary minerals for bone formation as xenograft don't resorb completely.

Xenografts undergoes deprotienaization by heating to eliminate the allergic reactions and risk of disease transmission .

The survival rate of implants with the use of xenografts as grating material is the same as implants using autogenous bone grafts .

Xenografts has the disadvantages of that there is a risk of cross contamination and possible development of immune reaction as there is no way to adequately screen them .

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with badly broken teeth in upper esthetic zone indicated for extraction, presence of at least 4 mm of bone beyond the root apex to guarantee implant primary stability, implant placement within the alveoli confines.
* Both sexes.
* No intraoral soft and hard tissue pathology.
* No systemic condition that contraindicate implant placement.

Exclusion Criteria:

* Presence of fenestrations or dehiscence of the residual bony Walls after extraction.
* Heavy smokers more than 20 cigarettes per day .(24)
* Patients with systemic disease that may affect normal healing.
* Psychiatric problems

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2020-06-10 (Actual); Study Completion 2020-06-10 (Actual)

PRIMARY OUTCOMES:
crestal bone loss | 4 month
  the amount of crestal bone loss will be measured using cone beam computed tomography

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt